CLINICAL TRIAL: NCT06288503
Title: A Double-blind, Randomised-controlled Trial Evaluating a Hydrolysed Rice Formula Compared to a Cow's Milk Protein-based Extensively Hydrolysed Formula in Infants with Cow's Milk Allergy
Brief Title: Hydrolysed Rice Formula Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRF2023
Record Dates: First submitted 2024-02-01; First posted 2024-03-01 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Hydrolysed rice protein formula
  Interventions: Other: Hydrolysed Rice Protein Formula
- Control (Active Comparator): Cow's milk based extensively hydrolysed formula
  Interventions: Other: Cow's Milk Based Extensively Hydrolysed Formula

INTERVENTIONS:
Other: Hydrolysed Rice Protein Formula — Infants randomised onto this arm will be taking the hydrolysed rice protein formula, with a minimum prescription of 30% of their energy requirements.
  Arms: Intervention
Other: Cow's Milk Based Extensively Hydrolysed Formula — Infants randomised onto this arm will be taking the control product, with a minimum prescription of 30% of their energy requirements.
  Arms: Control

SUMMARY:
This non-inferiority study aims to determine whether a hydrolysed rice protein formula is as effective as a cow's milk protein based extensively hydrolysed formula using a double-blind, randomised-controlled design over a 28-day intervention period followed by a 2-month follow-up period in infants 0-13 months of age presenting with symptoms/clinical history suggestive of cow's milk allergy. The primary outcome is growth, and secondary outcomes are gastrointestinal tolerance, and differences in intake, allergic symptoms, parental QOL, acceptability, dietary intake, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 0-13 months
* Presenting to primary or secondary care with symptoms/clinical history suggestive of CMA
* Will receive at least 30% of energy requirements from the study formula
* Written informed consent from parent/carer

Exclusion Criteria:

* Severe CMA (including anaphylaxis) and/or requiring an AAF
* Faltering growth (based on NICE guidelines36 - Appendix 1)
* Previous allergy to any study product ingredients (including whey hydrolysate and/or rice)
* Primary lactose intolerance
* Food Protein-Induced Enterocolitis Syndrome (FPIES)
* Exclusively breast fed
* Severe concurrent or chronic disease or genetic syndrome that may impact growth or other outcomes
* Severe hepatic or renal insufficiency
* Premature infants (born <37 weeks) with a corrected age of <4 weeks
* Requirement for any parenteral nutrition
* Participation in other clinical intervention studies within 1 month of recruitment
* Concern around the willingness/ability of the caregiver to comply with the study protocol and/or study requirements

Ages: 0 Months to 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Growth | Baseline to three months
  At Baseline (Day 1), End of Intervention (Day 31), and Follow-Up (Day 87) assessments, length and head circumference will be measured using standard measures to the nearest 0.1cm. Body weight (kg) will also be measured, where possible, by the investigating Dietitian/relevant HCP using standard methods to the nearest 0.1kg using a weighing scale without heavy clothing. These measures will be used to calculate z-scores (i.e., weight-for-length, weight, length, and head circumference; based on UK-WHO 2006 growth reference data for children 0-4 years old) and plotted on growth charts for centile measurement.

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Baseline to three months
  Gastrointestinal tolerance will be recorded by the parent/carer at Baseline Assessment and Baseline Days 1-3, where this period is undertaken by the patient), during the Intervention Period on Days 10, 17, 24, and 29-31, and during the 2-month Follow-Up period on Days 85-87. Tolerance will be recorded using a standardised GI tolerance questionnaire.
Stool frequency and consistency | Baseline to three months
  Stool frequency and consistency (Brussels Infant and Toddler Stool Scale) will be recorded by the parent/carer at Baseline on Days 1-3 (where applicable), as well as on during the Intervention Period on Days 10, 17, 24, and 29-31, and during the 2-month Follow-Up on Days 85-87.
Study Product Intake | Baseline to three months
  Intake of study product will be assessed daily throughout the Baseline and Intervention Periods by the parent/carer by recording how much feed was consumed. During the 2-month Follow-Up, intake of study product will be assessed for 3 days (Days 84-87). The daily minimum target intake amount prescribed by the investigating Dietitian/relevant HCP will be recorded at the start of the study, and any changes to this prescription will be noted.
Patient Orientated Scoring Atopic Dermatitis Symptoms (PO-SCORAD) | Baseline to three months
  A self-evaluation tool will be completed by the parent/carer on the day of the Baseline Assessment (Day 1), on Days 10 and 31 during the Intervention Period, and on Day 87 during the 2-month Follow-Up to give an indication of severity of atopic dermatitis (where present). This will involve tick box questions and a diagram of an infant for the parent/carer to highlight presence of dermatitis.
Patient Reported Atopic Symptoms | Baseline to three months
  The parent/carer will be asked to indicate their perception of the presence and severity of several common atopic symptoms for their child (wheezing, itchy/watery eyes, crying frequency, sneezing/runny/blocked nose, sleep quality) via 100mm visual analogue scales, with 100mm indicating more severe symptoms. These will be recorded on at Baseline Assessment (Day 1), on Day 3, Days 10, 17, 24, and 31 during the Intervention Period, and on Day 87 during the Follow-Up Period.
Cow's Milk Related Symptom Score | Baseline to three months
  Infants' stool pattern, the presence and intensity of crying and regurgitation, as well as skin and respiratory manifestations will be assessed via the CoMiSS™ tool by the investigating Dietitian/relevant HCP at the Baseline (Day 1), End of Intervention (Day 31), and Follow-Up (Day 87) Assessments. Total scores range from 0-33, with higher number indicating more severe symptoms of cow's milk allergy.
Food Allergy Quality of Life-Parental Burden (FAQL-PB) | Baseline to three months
  Parental measures of QOL (related to their child's allergy) will be assessed via a standardised validated questionnaire on the day of the Baseline Assessment (Day 1), on the final day of the Intervention Period (Day 31), and at the end of the Follow-Up Period (Day 87).
Acceptability of the Study Formula | Baseline to three months
  Feed acceptability (e.g., ease of use, liking) will be assessed at Baseline (Day 3, where applicable), during the Intervention Period on Days 10 and 31, and at the end of the Follow-Up period on Day 87, via a Likert-style questionnaire completed by the parent/carer (strongly disagree/disagree/don't know/agree/strongly agree)
Nutrient Intake (Energy, Protein, Micronutrients) | Baseline to three months
  Nutrient intake, including intake of all nutrition provided (including the study product, any other enteral feeding, foods, drinks etc.) will be recorded via a 24hr dietary recall conducted by the investigating Dietitian/relevant HCP at the Baseline (Day 1), Day 10, End of Intervention (Day 31), and Follow-Up (Day 87) Assessments. Dietary data will be inputted by the study team into nutritional software to estimate energy and macro- and micronutrient intakes.
Dietetic Goal | Baseline to three months
  A dietetic goal (e.g., improve tolerance, reduce atopic symptoms, maintain symptom control, maintain normal growth) will be set by the investigating Dietitian/relevant HCP at the Baseline Assessment (Day 1) for each infant. At the End of Intervention Assessment (Day 31), the investigating Dietitian/relevant HCP will assess and note if the dietetic goal was met (yes/no) and will set a dietetic goal for the Follow-Up Period. At the Follow-Up Assessment (Day 87), the investigating Dietitian/relevant HCP will assess and note if the dietetic goal was met (yes/no).
Overall Safety | Through study completion, an average of three months
  All adverse events will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Gloucestershire Royal NHS Trust, Gloucester, Gloucestershire
  - Bristol Royal Hospital for Children, Bristol, Somerset

IPD SHARING:
Plan to Share IPD: No